CLINICAL TRIAL: NCT06096038
Title: Administration of T Cells Expressing Chondroitin-Sulfate-Proteoglycan-4 Specific Chimeric Antigen Receptors (CAR) in Subjects With Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Autologous CAR-T Cells Targeting CSPG4 in Relapsed/Refractory HNSCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Bellicum Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2060-ATL; R01CA296807-01 (NIH)
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Cancer; Relapse; Recurrent; Refractory Cancer
Keywords: cellular therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Recurrence; Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chimeric Antigen Receptors (Experimental): blood will be collected to prepare the iC9.CAR-CSPG4 T cells. Disease-fighting T cells will be isolated and modified to prepare the iC9.CAR-CSPG4 T cells. In part 2, the iC9.CAR-CSPG4 T cells are given by infusion after completion of lymphodepletion chemotherapy.
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Cell Therapy

INTERVENTIONS:
Drug: Cyclophosphamide — cyclophosphamide 300 mg/meter square IV
  Other Names: Cycloblastin; Cytoxan; Endoxan; Neosar; Procytox; Revimmune
Drug: Fludarabine — fludarabine 30 mg/meter square IV × 3 days
  Other Names: Fludara; Fludarabine Phosphate
Biological: Cell Therapy — the autologous T lymphocyte chimeric antigen receptor cells against the CSPG4 antigen iC9-CAR.CSPG4 T cell infusion iC9-CAR.CSPG4 T cell infusion

SUMMARY:
The purpose of this study is to test the safety and tolerability of using a new treatment called autologous T lymphocyte chimeric antigen receptor cells against the CSPG4 antigen (iC9.CAR-CSPG4 T cells) in patients with head and neck cancer that came back after receiving standard therapy for this cancer. The iC9.CAR-CSPG4 treatment is experimental and has not been approved by the Food and Drug Administration.

How many (dose) of the iC9.CAR. CSPG4 T cells are safe to use in patients without causing too many side effects, and what is the maximum dose that could be tolerated will be investigated. The information collected from the study would help cancer patients in the future.

There are two parts to this study. In part 1, blood will be collected to prepare the iC9.CAR-CSPG4 T cells. Disease fighting T cells will be isolated and modified to prepare the iC9.CAR-CSPG4 T cells. In part 2, the iC9.CAR-CSPG4 T cells are given by infusion after completion of lymphodepletion chemotherapy.

The data from the dose escalation will be used to determine a recommended phase 2 dose (RP2D), which will be decided based on the maximum tolerated dose (MTD). Additionally, recommended phase 2 dose will be tested.

Eligible subjects will receive lymphodepletion chemotherapy standard followed by infusion of iC9-CAR.CSPG4 T cells. After treatment completion or discontinuation, subjects will be followed since involving gene transfer experiments.

ELIGIBILITY:
Inclusion Criteria:

Unless otherwise noted, subjects must meet all of the following criteria to participate in all phases of the study:

1. Written informed consent and HIPAA authorization for release of personal health information explained to, understood by and signed by the subject; subject given a copy of the informed consent form.
2. Age ≥ 18 years at the time of consent.
3. Karnofsky score of > 60%
4. Histologically or cytologically confirmed stage recurrent/metastatic squamous cell carcinoma of the head and neck as defined by American Joint Committee on Cancer (AJCC). This includes squamous cancer of: oral cavity, oropharynx, hypopharynx and larynx.

Exclusion Criteria:

1. Subject with a history or current severe progressive heart disease (congestive heart failure, coronary artery disease, uncontrolled arterial hypertension, uncontrolled arrhythmia, or myocardial infarction in the past 6 months.
2. Subject with a history of stroke or transient ischemic attack (TIA) within 12 months before procurement.
3. Subject with a history of severe immediate hypersensitivity reaction to cyclophosphamide or fludarabine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Toxicity: NCI-CTCAE | Up to 4 weeks
  Toxicity will be graded as the Number of participants with adverse events (AE)s
  AEs will be classified and graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Dose Limiting Toxicities (DLTs) is defined as at least possibly related to CAR.B7-H3T cell product administration.
Toxicity: Cytokine Release Syndrome (CRS) | Up to 4 weeks
  CRS will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) CRS Consensus Grading. Grade 1 - Mild: Fever ≥38^ o C, No hypotension, No hypoxia, Grade 2 - Moderate: Fever ≥38^ o C, Hypotension not requiring vasopressors, Hypoxia requiring low-flow nasal cannula (≤6 L/minute) or blow-by, Grade 3 - Severe: Fever ≥ 38^ o C, Hypotension requiring a vasopressor with or without vasopressin, Hypoxia requiring high-flow nasal cannula (>6 L/minute), facemask, nonrebreather mask, or Venturi mask, Grade 4 - Life-threatening: Fever ≥38^oC, Hypotension requiring multiple vasopressors (excluding vasopressin), Hypoxia requiring positive pressure (e.g. Continuous positive airway pressure, BiPAP, intubation, mechanical ventilation), Grade 5 - Death
Toxicity: Immune effector cell-associated neurotoxicity syndrome (ICANS) | Up to 4 weeks
  Neurotoxicity will be graded according to the Immune effector cell-associated neurotoxicity syndrome (ICANS) criteria.
  Immune effector cell-associated neurotoxicity syndrome (ICANS) symptoms will be graded according to the criteria outlined in the protocol on a scale from 1 (mild) to 4 (critical). Cytokine release syndrome (CRS) will be graded according to criteria outlined in the protocol on a scale from 1 (mild) to grade 5 (death).
Dose Limiting Toxicity | Up to 4 weeks
  An event will be considered a Dose limiting toxicity per NCI CTCAE version 5.0, the CRS Grading and ICANS grading criteria.
  * Grade 3-5 allergic reactions related to the CAR-T cell infusion.
  * A treatment-emergent Grade 3 CRS that does not improve to Grade 0-1 by 72 hours or Grade 4 CRS
  * Grade ≥3 ICANS that is unresponsive to the standard of care interventions and does not decrease to Grade ≤1 within 7 days or grade 4 ICANS of any duration that has evidence of cerebral edema and/or generalized convulsive status epilepticus.
  * Any treatment-emergent Grade 4 non-hematologic AE that does not resolve to Grade 2 within 7 days.
  * Any Grade 5 events are not due to the underlying malignancy.

SECONDARY OUTCOMES:
The recommended phase 2 dose (RP2D) of iC9-CAR.CSPG4 | Up to 4 weeks
  The recommended phase 2 dose (RP2D) for administration of iC9-CAR.CSPG4 T cells will be determined based on the modified 3+3 dose finding rule and the tolerability of iC9-CAR.CSPG4 T cells. tolerability of iC9-CAR.CSPG4 T cells will be assessed by NCI-CTCAE v5, ASTCT Consensus ICANS Grading, and CRS Grading Criteria.
Objective response rate | Up to 2 years
  The objective response rate will be assessed per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) and immune-related Response Evaluation Criteria in Solid Tumors (irRECIST).
  RECIST v1.1: Complete Response (CR) as Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; and Overall Response Rate (ORR) = CR + PR/total number of subjects.
  irRECIST: Complete Response (irCR), Disappearance of all lesions, no new lesions, lymph nodes < 10 mm in short axis; Partial Response (irPR), ≥30% decrease in the sum of target lesions and non-target lesions are irNN; Stable response (irSD), not meeting criteria for irCR, irPR, or irPD; Progressive Disease (irPD), ≥20% increase in tumor burden and minimum 5 mm absolute increase in compared to nadir.

OTHER OUTCOMES:
Progression Free Survival (PFS) | Up to 2 years
  PFS will be measured from the first day of lymphodepletion chemotherapy prior to iC9- CAR.CSPG4 T cell infusion to progression per RECIST 1.1 or death.
Overall Survival (OS) | Up to 2 years
  OS will be measured from the first day of lymphodepleting chemotherapy prior to iC9-CAR.CSPG4 T cell infusion to date of death for any cause.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the time from partial response (PR) or better to progressive disease (PD) per RECIST 1.1. and irRECIST.
Feasibility of iC9-CAR.CSPG4 T cell therapy | From cell procurement to 4 weeks after iC9-CAR.CSPG4 T cell infusion.
  Feasibility will be determined by measuring the percent of subjects procured that proceed with lymphodepletion followed by iC9-CAR.CSPG4 T cell infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Weiss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials